CLINICAL TRIAL: NCT02999282
Title: Rehabilitative Trial for the Recovery of Neurophysiological Parameters in Progranulin Mutation Carriers Through the Use of Transcranial Direct Current Stimulation (tDCS)
Brief Title: Rehabilitative Trial for the Rescue of Neurophysiological Parameters in Progranulin Deficient Subjects
Acronym: ReRescuePGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Associated Professor; MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NP2441
Record Dates: First submitted 2016-12-02; First posted 2016-12-21 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Frontotemporal Dementia; GRN Related Frontotemporal Dementia
Keywords: TMS; tDCS; Rehabilitation
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Presymptomatic real tDCS (Experimental): Asymptomatic subjects - 10 days anodal transcranial direct current stimulation
  Interventions: Device: Anodal transcranial direct current stimulation
- Presymptomatic sham tDCS (Sham Comparator): Asymptomatic subjects - 10 days sham transcranial direct current stimulation
  Interventions: Device: Sham transcranial direct current stimulation
- Symptomatic real tDCS (Experimental): Symptomatic patients - 10 days anodal transcranial direct current stimulation
  Interventions: Device: Anodal transcranial direct current stimulation
- Symptomatic sham tDCS (Sham Comparator): Symptomatic patients - 10 days sham transcranial direct current stimulation
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation — 10 sessions of anodal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Presymptomatic real tDCS; Symptomatic real tDCS
Device: Sham transcranial direct current stimulation — 10 sessions of sham transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Presymptomatic sham tDCS; Symptomatic sham tDCS

SUMMARY:
In this randomized, double-blind, sham-controlled study, the investigators will evaluate the effects of frontal and prefrontal anodal transcranial direct current stimulation (tDCS) on neurophysiological parameters of cortical connectivity, assessed by transcranial magnetic stimulation (TMS), in asymptomatic subjects bearing a pathogenic GRN mutation and in symptomatic patients with frontotemporal dementia.

DETAILED DESCRIPTION:
In this randomized, double-blind, sham-controlled study, the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation (tDCS) on neurophysiological parameters of cortical connectivity, assessed by transcranial magnetic stimulation (TMS), in asymptomatic subjects bearing a pathogenic GRN mutation and in symptomatic patients with frontotemporal dementia.

All patients will undergo genetic screening for progranulin mutations, a baseline neuropsychological and neurophysiological evaluation, including assessment of short interval intracortical inhibition, intracortical facilitation, short interval intracortical facilitation and long interval intracortical inhibition. Subjects will then be randomized in two groups, one receiving a 10 day (5 days/week for 2 weeks) treatment with anodal frontal and prefrontal anodal tDCS and the other receiving sham stimulation with identical parameters. After the intervention, patients will be reassessed with a neuropsychological and neurophysiological evaluation at 2 weeks, 1 month (only neurophysiological evaluation), 3 months and 6 month after treatment.

ELIGIBILITY:
Inclusion Criteria: presymptomatic carriers, symptomatic genetic FTD patients, symptomatic sporadic FTD patients.

* Presymptomatic carriers: defined as participants who are known carriers of a pathogenic mutation in the GRN gene, who do not fulfill current criteria for the behavioral variant FTD (bvFTD) (Rascovsky et al. 2011) or for the Primary Progressive Aphasias (PPA) (Gorno-Tempini et al. 2011). All subjects will be genotyped for known pathogenic mutations for FTD (GRN, C9orf72, MAPT, TDP-43) before participation.
* Symptomatic genetic FTD: defined as patients who are known carriers of pathogenic mutation in the GRN gene, fulfilling current clinical criteria for behavioral variant FTD (bvFTD) (Rascovsky et al. 2011) or the agrammatic variant of Primary Progressive Aphasia (avPPA) (Gorno-Tempini et al. 2011).
* Symptomatic sporadic FTD: defined as patients fulfilling current clinical criteria for behavioral variant FTD (bvFTD) (Rascovsky et al. 2011) or the agrammatic variant of Primary Progressive Aphasia (avPPA) (Gorno-Tempini et al. 2011), with a negative screening for pathogenic mutations in known FTD genes (GRN, C9orf72, MAPT, TDP-43). CSF analysis or amyloid PET imaging will be carried out to exclude focal variants of AD.

Exclusion Criteria:

* Cerebrovascular disorders, previous stroke, hydrocephalus, and intra-cranial mass documented by MRI.
* History of traumatic brain injury or other neurological diseases.
* Serious medical illness other than FTD
* History of seizures
* Pregnancy
* Metal implants in the head (except dental fillings)
* Electronic implants (i.e. pace-maker, implanted medical pump)
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in SICI measurements from Baseline | Baseline - 2 weeks
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on short interval intracortical inhibition (SICI)
Change in ICF measurements from Baseline | Baseline - 2 weeks
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on intracortical facilitation (ICF).

SECONDARY OUTCOMES:
Change in SICI measurements from Baseline | Baseline - 1 month - 3 months - 6 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on short interval intracortical inhibition (SICI)
Change in ICF measurements from Baseline | Baseline - 1 month - 3 months - 6 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on intracortical facilitation (ICF).
Change in LICI measurements from Baseline | Baseline - 1 month - 3 months - 6 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on long interval intracortical inhibition (LICI).
Change in SICF measurements from Baseline | Baseline - 1 month - 3 months - 6 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of frontal and prefrontal anodal transcranial magnetic stimulation on short interval intracortical facilitation (SICF).
Change in MMSE scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  The Mini Mental State Examination (MMMSE) is a 30-point questionnaire that is used to measure cognitive impairment.
Change in phonemic fluencies scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Produce as many words as possible beginning with a specified letter in 60 seconds
Change in semantic fluencies scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Produce as many words as possible from a category in 60 seconds
Change in digit span forward scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Participants hear a sequence of numerical digits and are tasked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered.
Change in digit span backward scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Participants hear a sequence of numerical digits and are tasked to recall the sequence correctly in reverse order, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered.
Change in camel and cactus test scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Evaluates associative semantic memory with 64 items presented for naming and word-picture matching.
Change in TMTA scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  The task requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper to examine cognitive processing speed.
Change in TMTB scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  The task requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper, alternating between numbers and letters, to examine executive functioning.
Change in Stroop test scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Measure a person's selective attention capacity and skills, as well as their processing speed ability.
Change in Symbol Digit test scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  It consists of digit-symbol pairs followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured.
Change in Block Design test scores from Baseline | Baseline - 2 weeks - 3 months - 6 months
  To evaluated spatial visualization ability and motor skills. The test-taker uses hand movements to rearrange blocks that have various color patterns on different sides to match a pattern. The items in a block design test are scored both by accuracy in matching the pattern and by speed in completing each item.
Change in The modified EkmanFaces Test from Baseline | Baseline - 2 weeks - 3 months - 6 months
  Each face is presented on a sheet with six labels of basic emotions below the photograph. The patient was required to respond verbally, deciding the label that best described the facial expression shown.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data, including outcome measure results, study protocol and statistical analysis plan, will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the study completion indefinitely.
Access Criteria: Reasonable request

REFERENCES:
- [Background] Benussi A, Cosseddu M, Filareto I, Dell'Era V, Archetti S, Sofia Cotelli M, Micheli A, Padovani A, Borroni B. Impaired long-term potentiation-like cortical plasticity in presymptomatic genetic frontotemporal dementia. Ann Neurol. 2016 Sep;80(3):472-6. doi: 10.1002/ana.24731. Epub 2016 Aug 10. PMID 27438089
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650